CLINICAL TRIAL: NCT07094282
Title: Prospective Assessment of Integrative Therapies for Neuromusculoskeletal Pain (PAIN)
Acronym: PAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Moss (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, David Moss, Principal Investigator/Doctor, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOMMC.2025.0019
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain
Keywords: integrative medicine
MeSH Terms: conditions — Chronic Pain | interventions — Acupuncture Therapy; Myofascial Release Therapy; Lasers; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Single group single site prospective cohort. Patients will act as their own control with pre-intervention scores.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrative Medicine (pre to post treatment) (Experimental): Patients will act as their own control with preintervention scores. The main integrative medicine intervention therapies include but may not be limited to acupuncture, myofascial therapies, microcurrent therapies, LASER therapy, extracorporeal shockwave therapy, and pulsed electromagnetic therapies.
  Interventions: Other: Acupuncture; Other: myofascial therapy; Other: microcurrent therapy; Other: LASER; Other: extracorporeal shockwave therapy; Other: Pulsed electromagnetic therapies; Other: Miscellaneous integrative medicine

INTERVENTIONS:
Other: Acupuncture — Integrative Medicine: Acupuncture treatment
Other: myofascial therapy — Integrative Medicine: myofascial therapy to include transverse abdominus teaching, rectus abdominus release, functional neuromyofascial techniques, cupping, gua sha, active needling.
Other: microcurrent therapy — Integrative Medicine: Microcurrent
Other: LASER — Integrative Medicine: LASER
Other: extracorporeal shockwave therapy — Integrative Medicine: Extracorporeal shockwave therapy
Other: Pulsed electromagnetic therapies — Integrative Medicine: Pulsed electromagnetic therapies
Other: Miscellaneous integrative medicine — other integrative medicine modalities

SUMMARY:
With vast numbers of active-duty members restricted from their specific duties or deemed unfit for deployment because of low back pain, both the mission of the Department of Defense and overall military workflow can be significantly impacted. More than restriction from duty or being barred from deployment, studies have shown musculoskeletal conditions were among the top reasons for medical disability retirement in the Army and Marine Corps (Niebuhr; Sikorski). Given the significant time, money, and resources invested in training these members, each day of inactivity or disability detrimentally affects the execution of the military's mission. Therefore, precise diagnosis and effective treatment modalities are paramount to foster healing and reduce recovery time.

From an operational standpoint, the United States Department of Defense (DoD) is specifically interested in using tailored integrative medicine modalities to manage chronic conditions encountered in the military health system. Not just chronic pain, but polytrauma and the triad of conditions it encompasses; traumatic brain injury and post-traumatic stress disorder combined with chronic pain (Madsen, Kim, Bedard). The DoD's goal is also to decrease opioid prescribing and the addiction and altered state associated with opioids.

AT the Nellis Integrative Medicine Clinic, physicians, a chiropractor, and nurses are engaged in the treatment of patients. All personnel are trained in the various modalities available in the clinics.

A variety of modalities are utilized in the clinic. This prospective study will evaluate the effectiveness of the many modalities used in the Integrative Medicine Clinic (such as acupuncture, myofascial therapies, microcurrent therapies, LASER therapy, extracorporeal shockwave therapy, and pulsed electromagnetic therapies).

Most patients receive treatments using multiple modalities. DoD goals align with our experiences in the Integrative Medicine Clinic at Mike O'Callaghan Military Medical Center. Many servicemembers and dependents in our clinic are trying to avoid surgery, or their pain medications - opioid or not - are no longer working. Additionally, many patients are trying to avoid Do Not Fly status caused by pharmacologic approaches. Patient experiences at our IMC also correlate with a study where 80% of people surveyed felt integrative medicine should be routinely offered at all MTFs (Ross). While our patients generally are not on opioids, we have anecdotally noted a reduction or cessation of opioids in several patients. The impacts of such a reduction in opioid usage for military readiness is clear (Madsen).

DETAILED DESCRIPTION:
All of the below items are research-related unless marked as 'standard of care'. Visits will vary depending on provider-decided treatments and will generally range from 30 minutes to 2 hours in length.

Self-reported pain intensity assessment.

Screening visit (1 hour):

* Obtain and document signed Informed Consent document and HIPAA Authorization
* Verify subject eligibility based on inclusion/exclusion criteria. Medical record will verify inclusion.
* -Record all medications including over the counter the subject is taking. Record morphine milligram equivalents (MME) for patients taking opioid medications. Collect basic demographic information to include phone number, email address, DoD ID, age, race, ethnicity, assigned sex at birth, weight (pounds), height (inches), and BMI, estimated annual income.
* Collect additional information to include:

  * Beneficiary Status (Active-Duty, Retired Active-Duty, dependent, Reservist)
  * rank (if applicable),
  * employment status and description (full time, part time, unemployed, retired, homemaker) number of deployments (if applicable), Marital status (Married, Domestic Partners, Divorced, Widow/er, separated, single/never married)
  * education (military training; high school/GED; some college; 2 year college; 4 year college; some graduate work; completed master's or professional degree; completed Ph.D., law degree, MD, similar advanced professional degree)
* Patient History, was there a precipitating injury, location of pain (neck, thoracic, or lumbar), history of surgery and type of surgery, any history of pain management interventions (injections, ablations, etc) especially related to the subject's chronic axial spine pain
* Other therapies for their condition currently receiving or in the last 3 months (ie chiropractic, physical therapy, pain management etc) Randomization: Subjects will not be randomized as this is a single armed cohort study. Subjects will be assigned a unique study code in sequential order beginning with 001.

SURVEY RELATED VISITS

Visit 1 (week 0 can be the same day as screening visit) (30 minutes) (In-person or Virtual):

BASELINE

* Subject will fill out the following Standard of Care Patient Questionnaires:
* PROMIS Physical Function Form 6b
* 6 questions evaluating physical function
* DVPRS 0-10 Scale
* pain assessment tool using numerical rating scale enhances by functional word descriptors, color coding, and pictorial facial expressions
* PEG
* Assesses pain intensity and interference
* Patient Health Questionnaire 2-item (PHQ-2)
* Measures depressed mood and anhedonia over past 2 weeks
* Survey is extended to a 9-item PHQ-9 only for subjects scoring 3 or higher on the PHQ-2
* Generalized Anxiety Disorder 2-item (GAD-2)
* Screening tool for generalized anxiety disorder
* Survey is extended to a 7-item GAD-7 only for subjects scoring 3 or higher on the GAD-2
* Pain Catastrophizing Scale
* Quantifies pain experience (rumination, magnification, and helplessness)
* Pittsburgh Sleep Quality Index
* Dallas Pain Questionnaire
* 16 item quality of life questionnaire assessing multiple domains
* Patient receives treatment preferably same day, but within 72 hours
* Scores may be pulled from patient Electronic Medical Record

Visit 2 (Week 4) (60 minutes) (In-person or Virtual) Research coordinator with record morphine milligram equivalents (MME) for patients taking opioid medications.

* Subject will complete the following Standard of Care Patient Questionnaires:
* PEG
* PHQ-2 or PHQ-9 (PHQ-2 score > 2)
* GAD-2 or GAD-7 (GAD-2 score > 2)
* Pain Catastrophizing Scale
* Pittsburgh Sleep Quality Index
* DVPRS 0-10 Scale
* PROMIS Physical Function Form 6b
* Dallas Pain Questionnaire
* Scores may be pulled from patient Electronic Medical Record

Visit 3 (Week 8) (60 Minutes) (In-person or Virtual) Research coordinator with record morphine milligram equivalents (MME) for patients taking opioid medications.

* Subject will complete the following Standard of Care Patient Questionnaires:
* PEG
* PHQ-2 or PHQ-9 (PHQ-2 score > 2)
* GAD-2 or GAD-7 (GAD-2 score > 2)
* Pain Catastrophizing Scale
* Pittsburgh Sleep Quality Index
* DVPRS 0-10 Scale
* PROMIS Physical Function Form 6b
* Dallas Pain Questionnaire
* Scores may be pulled from patient Electronic Medical Record

Visit 4 (Week 12) (60 Minutes) (In-person or Virtual) Research coordinator with record morphine milligram equivalents (MME) for patients taking opioid medications.

* Subject will complete the following Standard of Care Patient Questionnaires:
* PEG
* PHQ-2 or PHQ-9 (PHQ-2 score > 2)
* GAD-2 or GAD-7 (GAD-2 score > 2)
* Pain Catastrophizing Scale
* Pittsburgh Sleep Quality Index
* DVPRS 0-10 Scale
* PROMIS Physical Function Form 6b
* Dallas Pain Questionnaire
* Patient receives treatment at provider discretion
* Scores may be pulled from patient Electronic Medical Record

Visit 5 (Week 16) (60 minutes) (In-person or Virtual) Research coordinator with record morphine milligram equivalents (MME) for patients taking opioid medications.

* Subject will complete the following Standard of Care Patient Questionnaires:
* PEG
* PHQ-2 or PHQ-9 (PHQ-2 score > 2)
* GAD-2 or GAD-7 (GAD-2 score > 2)
* Pain Catastrophizing Scale
* Pittsburgh Sleep Quality Index
* DVPRS 0-10 Scale
* PROMIS Physical Function Form 6b
* Dallas Pain Questionnaire
* Scores may be pulled from patient Electronic Medical Record

Visit 6 (Week 20) (60 minutes) (In-person or Virtual) Research coordinator with record morphine milligram equivalents (MME) for patients taking opioid medications.

* Subject will complete the following Standard of Care Patient Questionnaires:
* PEG
* PHQ-2 or PHQ-9 (PHQ-2 score > 2)
* GAD-2 or GAD-7 (GAD-2 score > 2)
* Pain Catastrophizing Scale
* Pittsburgh Sleep Quality Index
* DVPRS 0-10 Scale
* PROMIS Physical Function Form 6b
* Dallas Pain Questionnaire
* Scores may be pulled from patient Electronic Medical Record

Visit 7 (Week 24) (60 minutes) (In-person or Virtual) Research coordinator with record morphine milligram equivalents (MME) for patients taking opioid medications.

* Subject will complete the following Standard of Care Patient Questionnaires:
* PEG
* PHQ-2 or PHQ-9 (PHQ-2 score > 2)
* GAD-2 or GAD-7 (GAD-2 score > 2)
* Pain Catastrophizing Scale
* Pittsburgh Sleep Quality Index
* DVPRS 0-10 Scale
* PROMIS Physical Function Form 6b
* Dallas Pain Questionnaire
* Scores may be pulled from patient Electronic Medical Record

Visit 8 (Week 28) (60 minutes) (In-person or Virtual) Research coordinator with record morphine milligram equivalents (MME) for patients taking opioid medications.

* Subject will complete the following Standard of Care Patient Questionnaires:
* PEG
* PHQ-2 or PHQ-9 (PHQ-2 score > 2)
* GAD-2 or GAD-7 (GAD-2 score > 2)
* Pain Catastrophizing Scale
* Pittsburgh Sleep Quality Index
* DVPRS 0-10 Scale
* PROMIS Physical Function Form 6b
* Dallas Pain Questionnaire
* Scores may be pulled from patient Electronic Medical Record
* Treatment Helpfulness Questionnaire
* Active duty members will be asked if duty, fitness or mobility restrictions were lifted during the study period

TREATMENT VISITS Treatments given in Integrative Medicine Clinic will be at provider discretion. Subjects will attend a minimum of 3 visits then additional treatment sessions will be at provider discretion as well.

The following semi structured clinical algorithm will be used by providers in the clinic.

Visit 1:

1. Initial interview with focus on whole person
2. Microcurrent standard protocols (Standard concussion protocol, Spinal Cord long)
3. Myofascial work to include transverse abdominus teaching, rectus abdominus release, other myofascial, time permitting or as needed
4. Optional Loan of microcurrent box with protocols at physician discretion
5. Optional loan of avazzia or alpha stim at physician discretion
6. Home Exercise Program handout (HEP2go)

   Visit 2:
7. Assess effect of prior myofascial work
8. Re-education of TA activation, additional myofascial work as needed (including lower trap and

   /or glut med activation)
9. Assess effect of Microcurrent
10. Optional Loan of microcurrent box with protocols at physician discretion
11. Optional loan of avazzia or alpha stim at physician discretion
12. create plan for visit 3 (this could include additional myofascial work, shock wave therapy, acupuncture/dry needling, avazzia or alpha stim)

    Visits 3 through final:
13. Continue treatment with any or all of the following modalities

a. Myofascial treatments (functional neuromyofascial techniques [FNT], cupping, gua sha, active needling) b. Frequency Specific Microcurrent (FSM) c. Avazzia d. Extracorporeal shock wave therapy (ESWT) e. Acupuncture/dry needling f. Alpha stim (cranio-electric stimulation) Coordinators will monitor subject visits either in-person post each visit or by accessing the EMR post each visit to record visit details. Visit Details to Record

* Visit Number (1-10, >10)
* ICD-10 codes
* Examples
* M54.2 Cervicalgia
* M54.5 Low Back Pain
* M79.7 Fibromyalgia
* Z73.3 PTSD*
* M54.9 Dorsalgia, unspecified
* F41.9 Anxiety
* M25.51 Shoulder Pain
* M54.6 Thoracic Spinal Pain
* M72.2 Plantar Fasciitis
* L90.5 Scar Conditions and Fibrosis of Skin
* Modalities Used
* Examples
* Myofascial modalities (FNT, cupping, scraping/gua sha, active needling)
* FSM
* Avazzia
* Acupuncture
* Dry needling
* Alpha Stim
* ESWT

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Active Duty and DoD Beneficiaries (i.e. former military, spouse, dependent child) aged 18 or older referred to the Nellis Integrative Medicine Clinic chronic back or neck pain
* Pain Chronicity Threshold (pain score ≥4/10 documented in EMR or reported by patient at least 2 times in one year and at least 30 days apart).

Exclusion Criteria:

* Enrolled in other pain management program (e.g. pain management, PT

  /OT)
* Anticipated Change of station, deployment, retirement from military service, separation from active or reserve military service (includes national guard) or plan to discontinue enrollment at MOMMC in <6 months
* Planned surgery during the study period
* Pregnancy
* <3 months post-partum
* Hypermobility disorders such as Ehlers Danlos
* Active cancer (cancer in remission is not an exclusion)
* Implanted electrical devices that cannot be turned off (ie pacemaker); implanted stimulators or pumps that can be turned off are not exclusionary
* Injury or surgery within the last 6 weeks
* Dementia
* Delirium
* Inability to make medical decisions or understand treatment plan as decided upon by principle or associate investigators
* Undergoing medical evaluation board
* Currently in the process of establishing or appealing VA disability rating, or planning to do so within the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Dallas Pain Questionnaire | baseline (pre-treatment) through study period (visit 1, week 0) (visit 2, week 4) (visit 3, week 8) (visit 4, week 12) (visit 5, week 16) (visit 6, week 20) (visit 4, week 24) (visit 8, week 28)
  16 item quality of life questionnaire assessing multiple domains
PROMIS physical function form 6b | baseline (pre-treatment) through study period (visit 1, week 0) (visit 2, week 4) (visit 3, week 8) (visit 4, week 12) (visit 5, week 16) (visit 6, week 20) (visit 4, week 24) (visit 8, week 28)
  6 questions evaluating physical function
Defense and Veterans Pain Rating Scale | baseline (pre-treatment) through study period (visit 1, week 0) (visit 2, week 4) (visit 3, week 8) (visit 4, week 12) (visit 5, week 16) (visit 6, week 20) (visit 4, week 24) (visit 8, week 28)
  pain assessment tool using numerical rating scale enhanced by functional word descriptors, color coding, and pictorial facial expressions
PEG (pain average, enjoyment of life, and general activity) | baseline (pre-treatment) through study period (visit 1, week 0) (visit 2, week 4) (visit 3, week 8) (visit 4, week 12) (visit 5, week 16) (visit 6, week 20) (visit 4, week 24) (visit 8, week 28)
  assesses pain intensity and interference
Patient Health Questionnaire 2-item (PHQ-2) | baseline (pre-treatment) through study period (visit 1, week 0) (visit 2, week 4) (visit 3, week 8) (visit 4, week 12) (visit 5, week 16) (visit 6, week 20) (visit 4, week 24) (visit 8, week 28)
  measures depressed mood and anhedonia over past 2 weeks
Patient health questionnaire 9-item | baseline (pre-treatment) through study period (visit 1, week 0) (visit 2, week 4) (visit 3, week 8) (visit 4, week 12) (visit 5, week 16) (visit 6, week 20) (visit 4, week 24) (visit 8, week 28)
  measures more detailed depressed mood and anhedonia if patient scores 3 or higher on phq-2
Generalized Anxiety Disorder 2-item | baseline (pre-treatment) through study period (visit 1, week 0) (visit 2, week 4) (visit 3, week 8) (visit 4, week 12) (visit 5, week 16) (visit 6, week 20) (visit 4, week 24) (visit 8, week 28)
  screening tool for generalized anxiety disorder
Generalized Anxiety Disorder 7-item | baseline (pre-treatment) through study period (visit 1, week 0) (visit 2, week 4) (visit 3, week 8) (visit 4, week 12) (visit 5, week 16) (visit 6, week 20) (visit 4, week 24) (visit 8, week 28)
  extended screening tool for generalized anxiety disorder to use if subjects score 3 or higher on GAD-2
Pain Catastrophizing Scale | baseline (pre-treatment) through study period (visit 1, week 0) (visit 2, week 4) (visit 3, week 8) (visit 4, week 12) (visit 5, week 16) (visit 6, week 20) (visit 4, week 24) (visit 8, week 28)
  quantifies pain experience (rumination, magnification, and helplessness)
Pittsburgh Sleep Quality Index | baseline (pre-treatment) through study period (visit 1, week 0) (visit 2, week 4) (visit 3, week 8) (visit 4, week 12) (visit 5, week 16) (visit 6, week 20) (visit 4, week 24) (visit 8, week 28)
  Self-report questionnaire that assesses sleep quality over a one-month time interval. The global score ranges from 0 to 21. Higher scores indicate poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic and clinical data will be acquired from 125 participants. All data will be de-identified prior to receipt by the repository, but the information needed to generate a global unique identifier for the NLM Data Archive (NDA) (clinicaltrials.gov) will be collected for each subject. Sufficient data from this project will be preserved to enable sharing via NDA data of sufficient quality to validate and replicate research findings described in the Aims. NLM requires data measured from human subjects to be shared using the NDA. Demographic data, clinical data, data collection tools and study protocols will be made available in the NDA.
Supporting Information: Study Protocol, ICF
Time Frame: All data will be deposited to clinicaltrials.gov starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates.
Access Criteria: Data will be findable for the research community through the NDA Collection that will be established when this application is funded. For all publications, an NDA study will be created. Each of those studies is assigned a digital object identifier (DOI). This data DOI will be referenced in the publication to allow the research community easy access to the exact data used in the publication.
  The research community will have access to data when the award ends. As required by NDA, studies will also be created that contain the data used for every publication. Those studies will be shared when the pre-print is available. NDA studies have digital object identifiers (DOI) to aid in findability. We will include that DOI in relevant publications. NDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now.